CLINICAL TRIAL: NCT04892290
Title: Effectiveness of Sphenopalatine Ganglion Block on Postdural Puncture Headache Treatment: A Retrospective Observational Study
Brief Title: Sphenopalatine Ganglion Block for Postdural Puncture Headache
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Burak Kaya, Anesthesiology and Reanimation Specialist, MD, Sakarya University
Other Study IDs: 71522473/050.01.04
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Postdural Puncture Headache
Keywords: Sphenopalatine Ganglion Block; Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Conservative Treatment; Sphenopalatine Ganglion Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group C: Postdural puncture headache patients treated with Conservative treatment
  Interventions: Other: Conservative Treatment for Postdural Puncture Headache
- Group SGB: Postdural puncture headache patients treated with Sphenopalatine Ganglion Block and conservative treatment
  Interventions: Other: Conservative Treatment for Postdural Puncture Headache

INTERVENTIONS:
Other: Conservative Treatment for Postdural Puncture Headache — The patients in Group C were given continuous bed rest in the supine position, 3000 mL daily hydration, 6 mg kg-1 aminophylline , 2 g day-1 paracetamol and 65 mg day-1 caffeine as conservative treatment. Topical SGB was applied to patients in Group SGB in addition to conservative treatment.
  Other Names: Sphenopalatine Ganglion Block

SUMMARY:
Background: Postdural puncture headache (PDPH), which is one of the complications of spinal anesthesia, is a condition that negatively affects the quality of life of patients, causes late mobilization and prolonged hospital stay. Sphenopalatine ganglion block (SGB) has created a minimally invasive, easy, and safe treatment alternative.

Objective: Evaluating the effectiveness of topical SGB on PDPH treatment. Design: Retrospective observational study Setting: Single center tertiary level of care hospital study. The files of PDPH patients between Jan 2018 and Jan 2020 were scanned.

Patients: PDPH patients aged 18-65 are included and any patients with primary/secondary headache history are excluded.

Main outcome measures: Patients were divided into 2 groups. The group that given only conservative treatment was named as Group C, and the group of patients who had additionally been applied SGB was named as Group SGB. Headache severity was measured with Visual Analogue Scale (VAS) at the 1st,3rd, 12th and 24th hours of the treatment, in supine and upright position.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years-old
* not having any headache diagnosis (G44 and subgroup according to the International Classification of Diseases-10 classification),
* developed PDPH according to the International Headaches Classification after the neuraxial procedure

Exclusion Criteria:

* history of primary headaches such as migraine, cluster type, tension type
* secondary headache such as preeclampsia / eclampsia, cerebral venous thrombosis, stroke, ruptured aneurysm, hypertensive encephalopathy, pituitary apoplexy, meningitis and subarachnoid hemorrhage
* any local or systemic infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postdural Puncture Headache patients
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Headache in Supine Position | 1st, 3rd, 12th and 24th hours of follow-up
  Headache severity changes with Visual Analogue Scale (VAS, 0-10, 0: no pain, 10:worst pain)

SECONDARY OUTCOMES:
Headache in Prone Position | 1st, 3rd, 12th and 24th hours of follow-up
  Headache severity changes with Visual Analogue Scale (VAS, 0-10, 0: no pain, 10:worst pain)
Successfully treated patients ratio | 24th hour of follow-up
  At the 24th hour of their follow-up, all patients with a VAS>3 (Visual Analogue Scale) headache in an upright position are considered as unsuccessful treatment and are directed to the epidural blood patch procedure. Both groups will be compared with successfully treated patients ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Kaya, MD, Principal Investigator — Sakarya University; Serbülent Gökhan Beyaz, Prof MD, Study Chair — Istinye University; Ayça Taş Tuna, As Prof MD, Study Chair — Sakarya University; Havva Kocayiğit, MD, Study Chair — Sakarya University
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Database